CLINICAL TRIAL: NCT01314729
Title: Clinical and Radiographic Comparison and Evaluation of Two Types of Lingual Fixed Retainers on the Health of Periodontium
Brief Title: Comparison of the Effect of Two Types of Fixed Retainers on the Health of the Gums
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Shiraz Dental School, Orthodontic Research Center (Unknown)
Responsible Party: Orthodontic Research Cneter, Shiraz Dental School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 8901372055shirazUMS
Record Dates: First submitted 2011-03-07; First posted 2011-03-14 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-02

CONDITIONS: Health of Periodontium
Keywords: Orthodontic fixed retainer; fiber-reinforced-composite retainer; composite-wire retainer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fiber-reinforced-composite retainer (Active Comparator)
  Interventions: Device: Fiber-reinforced-composite retainer
- composite-wire retainer (Active Comparator)
  Interventions: Device: Composite-wire retainer

INTERVENTIONS:
Device: Fiber-reinforced-composite retainer — this type of retainer is placed on the lingual surface of teeth from canine to canine just before the completion of orthodontic treatment
  Arms: Fiber-reinforced-composite retainer
Device: Composite-wire retainer — this type of retainer is placed on the lingual surface of teeth from canine to canine just before the completion of orthodontic treatment to prevent treatment relapse
  Arms: composite-wire retainer

SUMMARY:
Different types of retainers have been used to assure the stability of orthodontic treatment. The aim of this study is clinical and radiographic comparison and evaluation of two common types of lingual fixed retainers on the health of periodontium.

The participants in this study will be examined both clinically and radiographically just after the completion of orthodontic treatment and after a 6-month-period.

The results of the study will be analyzed with Mann-whitney and independent t-test.

ELIGIBILITY:
Inclusion Criteria:

1. The patient who have completed orthodontic treatment
2. The patients should be healthy with no systemic disease at the time
3. In clinical examination no apparent periodontal disease or inflammation should be present
4. Patients who have complete permanent dentition (3rd molar eruption is not required)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Measuring periodontal status through clinical examination | approximately 20 months
  for each participant, the examination is carried out right after the completion of orthodontic treatment and after a 6-month-period
measuring PDL width in periapical radiographs | approximately 20 months
  for each participant, the examination is carried out right after the completion of orthodontic treatment and after a 6-month-period

SECONDARY OUTCOMES:
Assessing periodontial status with Gingival Index | approximately 20 months
  A gingival Index score will be assigned to each patient upon completion of orthodontic treatment and after a 6-month-period
assessing periodontal status using Plaque Index | approximately 20 months
  A plaque Index score will be assigned to each patient upon completion of orthodontic treatment and after a 6-month-period
assessing periodontal status using Calculus Index | approximately 20 months
  A Calculus Index score will be assigned to each patient upon completion of orthodontic treatment and after a 6-month-period
assessing periodontal status using Bleeding on probing | approximately 20 months
  Each patient will be examined for bleeding on probing upon completion of orthodontic treatment and after a 6-month-period

CONTACTS AND LOCATIONS:
Overall Officials: Morteza Oshagh, Associate professor, Principal Investigator — Shiraz Dental School; Sepideh Torkan, resident, Principal Investigator — Shiraz Dental School
Locations (1):
- Shiraz Dental School, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Torkan S, Oshagh M, Khojastepour L, Shahidi S, Heidari S. Clinical and radiographic comparison of the effects of two types of fixed retainers on periodontium - a randomized clinical trial. Prog Orthod. 2014 Aug 27;15(1):47. doi: 10.1186/s40510-014-0047-8. PMID 25162332